CLINICAL TRIAL: NCT07087015
Title: Efficacy of Cervical Sympathetic Blocks for Post-traumatic Stress Disorder: a Randomized Control Trial
Brief Title: Efficacy of Cervical Sympathetic Blocks for PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Maria Bombardieri, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81697
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: cervical sympathetic nerve bock; regional anesthesia; neuromodulation; sympathetic blockade
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Twenty patients will be enrolled, with 10 patients allocated to each study arm (treatment and control).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (CSB) (Experimental): Patients will receive an ultrasound guided cervical sympathetic block. The block procedure consists of the deposition of local anesthetic under ultrasound guidance at the level of the cervical sympathetic ganglia.
  Interventions: Procedure: Cervical sympathetic nerve block; Drug: Ropivacaine
- Control group (Sham Comparator): Patients will receive a subcutaneous sham injection with saline. Ultrasound imaging will be used to simulate the guidance process as in the active procedure, maintaining consistency in the procedural experience.
  Interventions: Procedure: Subcutaneous sham injection; Drug: Normal Saline

INTERVENTIONS:
Procedure: Cervical sympathetic nerve block — Patients will receive a CSB.
  Arms: Intervention Group (CSB)
Procedure: Subcutaneous sham injection — Patients will receive a subcutaneous sham injection of saline.
  Arms: Control group
Drug: Ropivacaine — The CSB group will receive ropivacaine 0.5% 10ml.
  Arms: Intervention Group (CSB)
Drug: Normal Saline — The control group will receive 3 ml of normal saline in the sham injection.
  Arms: Control group

SUMMARY:
Millions of people suffer from anxiety disorders, including posttraumatic stress disorder (PTSD)-a condition that can profoundly disrupt daily life. Although treatments like therapy and medication help many, there is still a major need for more effective and faster-acting options. In recent studies, a procedure called cervical sympathetic block (CSB)-an injection near a nerve cluster in the neck-has shown promise in reducing PTSD symptoms, as measured by standardized tools like the CAPS (Clinician-Administered PTSD Scale). In this study, the investigators will conduct a double-blind, randomized controlled trial comparing CSB to a sham (placebo) injection in patients with PTSD. The investigators will assess changes in PTSD symptoms and also monitor physiological markers (like pupil response, temperature, and heart rate variability) to better understand how the treatment works and to improve the precision of future therapies.

DETAILED DESCRIPTION:
The investigators aim to determine whether cervical sympathetic blocks (CSBs) can reduce symptoms of posttraumatic stress disorder (PTSD). If effective, this approach could offer a rapid, legal, and scalable intervention for mental health conditions, in contrast with emerging psychedelic therapies. This research has the potential to transform treatment practices for PTSD and related disorders by providing a controlled, procedure-based option that modulates the autonomic nervous system. In addition to assessing symptom relief, the study will explore physiologic markers of sympathetic modulation, which may help identify objective indicators of treatment success. This could deepen our understanding of the neural mechanisms underlying PTSD and mental health more broadly, with implications for neuroscience, psychology, and clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age, inclusive, at screen.
2. Able to read, understand, and provide written informed consent in English prior to screening, and likely to comply with study procedures and communicate effectively with study personnel regarding adverse events or other clinically important information.
3. Diagnosed with PTSD prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition. The diagnosis of PTSD will be made by a trained study staff member and supported by the Structured Clinical Interview for DSM Disorders (SCID).
4. Meet the threshold of CAPS-5 score of >20 during screening.
5. Concurrent psychotherapy will be allowed if the type (e.g., supportive, cognitive behavioral, insight-oriented, et al) and frequency (e.g., weekly or monthly) of the therapy has been stable for at least 4 weeks prior to screening and if the type and frequency of the therapy is expected to remain stable during the course of the subject's participation in the study.
6. Concurrent antidepressant therapy (e.g. SSRI or SNRI) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.
7. In sufficiently good health to proceed with a low-risk elective procedure, characterized using the American Society of Anesthesiologists (ASA) physical status classification system as Class I, II, or III.

ASA Class III participants whose functional impairment is directly related to a psychiatric diagnosis (depression, anxiety or PTSD) will be included.

Exclusion Criteria:

* Allergy to local anesthetics
* Severe coagulopathy
* Female that is pregnant or breastfeeding.
* Female with a positive pregnancy test at screening or baseline.
* Total CAPS-5 score £20 at screening.
* Current diagnosis of a Substance Use Disorder (SUD; Abuse or Dependence, as defined by DSM-V) rated "moderate" or "severe" per criteria of the SCID, or Alcohol Use Disorder rated "moderate" or "severe" per SCID criteria. The following categories of SUD will NOT be excluded: nicotine dependence; alcohol or substance use disorder rated "mild"; alcohol or substance use disorder of any severity in remission, either early (3-12 months) or sustained (>12 months) time frames.
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Specific Phobia, or Bipolar II Disorder (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more)
* History of schizophrenia or schizoaffective disorders, or a psychotic disorder as defined by SCID interview.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their PTSD or has been predominant to their PTSD at any time within six months prior to screening.
* In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of his/her participation in the study.
* A neurological disorder including:

  1. Has dementia, delirium, amnestic, or any other cognitive disorder
  2. Encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation
  3. Any other disease/accident/intervention associated with significant injury to or malfunction of the central nervous system with ongoing clinically significant sequelae, or in the view of the investigator poses a risk for participation in this study.
* A cardiovascular disorder including:

  1. Uncontrolled hypertension
  2. Congestive heart failure NYHA Criteria >Stage 2
  3. Atrial fibrillation or resting heart rate <50 or >105 beats per minute at screening or randomization
  4. Any clinically significant conduction abnormalities (eg 2nd degree AV nodal block or left bundle branch block)
  5. QTcF (Fridericia-corrected) >= 450 msec at screening or randomization
  6. Any cardiovascular disorder that would merit categorization of patient as ASA Class III or higher
* A pulmonary/respiratory disorder including:

  1. Diagnosed Obstructive Sleep Apnea or STOPBANG score of 5 or higher
  2. History of difficult airway in surgical setting
  3. Any pulmonary / respiratory disorder that would merit categorization of patient as ASA Class III or higher
* Clinically significant liver disease, determined by LFTs within the past 6 months.
* Clinically significant kidney disease determined by GFR (<40 mL/min, Cockcroft-Gault Equation)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS-5) scores | Baseline (1 month before the block), 30 and 90 days post-block.
  CAPS-5 score is used to establish severity of PTSD. It is a 30-item structured interview that assesses the 20 DSM-5 PTSD symptoms, as well as associated features, the onset and duration of symptoms, global severity, symptom impact, improvement in symptoms, and a validity check. The resulting values range from 0 to 80, with the higher scores indicating worse PTSD symptom severity.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) scores | Baseline (1 month before the block), then 7, 14, 30 and 90 days post-block
  PCL-5 is used to establish severity of self-rated symptoms of PTSD. It is a 20-item self-report measure that assesses the 20 DSM-5 PTSD symptoms. The resulting valuea range from 0 to 80, with the higher scores indicating worse PTSD symptom severity.
Patient Health Questionnaire-9 (PHQ-9) | 2 weeks before the block and 2 weeks post-block
  A 9-item, self-administered instrument used to screen for the presence and severity of depression. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 27. Higher scores indicate greater depressive symptom severity.
State and Trait Anxiety Scale (STAI) | 2 weeks before the block and 2 weeks post-block
  A 40-item self-report questionnaire designed to assess two types of anxiety: state anxiety (temporary condition in response to specific situations) and trait anxiety (general tendency to respond with anxiety). Each subscale (20 items each) is scored on a 4-point Likert scale, with higher scores indicating greater anxiety.
Generalized Anxiety Disorder scale (GAD-7) | 2 weeks before the block and 2 weeks post-block
  A 7-item self-report questionnaire used to assess the severity of generalized anxiety symptoms over the past two weeks. Each item is scored from 0 ("not at all") to 3 ("nearly every day"), yielding a total score ranging from 0 to 21. Higher scores indicate greater levels of anxiety.
Positive and Negative Affect Schedule (PANAS) | 2 weeks before the block and 2 weeks post-block
  A 20-item self-report questionnaire that measures two distinct dimensions of affect: Positive Affect (PA) and Negative Affect (NA). Respondents rate the extent to which they have experienced various emotions over a specified time frame using a 5-point Likert scale (1 = very slightly or not at all; 5 = extremely). Each subscale consists of 10 items, with higher scores indicating greater positive or negative affect.
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks before the block and 2 weeks post-block
  A self-rated questionnaire that assesses sleep quality and disturbances over a 1-month period. It consists of 19 items generating seven component scores (e.g., sleep latency, duration, disturbances), which are summed to yield a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality.
The Satisfaction With Life Scale | 2 weeks before the block and 2 weeks post-block
  A 5-item self-report instrument designed to assess global cognitive judgments of one's overall life satisfaction. Each item is rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), producing a total score ranging from 5 to 35. Higher scores indicate greater life satisfaction.
Scales of Psychological Well-Being | 2 weeks before the block and 2 weeks post-block
  A multidimensional self-report instrument designed to assess six key aspects of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Versions range from 18 to 84 items, with each dimension measured via Likert-scale items. Higher scores reflect greater well-being in each domain.
Peace of Mind Scale | 2 weeks before the block and 2 weeks post-block
  A brief self-report measure assessing an individual's inner peace and emotional calmness. The scale typically consists of 5 items rated on a 5-point Likert scale (1 = not at all; 5 = extremely true), with higher scores indicating a greater sense of peace and psychological stability.
The Emotion Regulation Questionnaire Short Form | 2 weeks before the block and 2 weeks post-block
  A 6-item self-report instrument that assesses two emotion regulation strategies: cognitive reappraisal (4 items) and expressive suppression (2 items). Each item is rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with higher scores indicating greater use of the respective strategy.
Harmony in Life Scale | 2 weeks before the block and 2 weeks post-block
  A 5-item self-report measure that assesses an individual's perceived harmony and balance in life. Items are rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with higher scores indicating greater harmony in life.
The Perth Alexithymia Questionnaire Short Form | 2 weeks before the block and 2 weeks post-block
  A 24-item self-report questionnaire designed to assess alexithymia, characterized by difficulties in identifying, describing, and processing emotions. The PAQ measures both general alexithymia and its specific facets across different emotional valences (positive and negative). Items are rated on a 7-point Likert scale, with higher scores indicating greater alexithymic traits.
Stanford Expectations of Treatment Scale (SETS) | 2 weeks before the block and 2 weeks post-block
  A brief self-report measure assessing patients' positive and negative expectations regarding treatment outcomes. The scale consists of 10 items rated on a 5-point Likert scale, capturing the extent of optimism or pessimism about the effectiveness of a given treatment. Higher scores reflect stronger positive expectations.
Columbia Suicidality Severity Rating Scale (CSSRS) Short Screen | 3 weeks before the block and days 1, 7, 14, 30, 90 post-block
  A brief clinician- or self-administered screening tool designed to assess the severity and immediacy of suicidal ideation and behavior. The short screen includes key items to quickly identify individuals at risk by evaluating recent suicidal thoughts, plans, and attempts. While the full C-SSRS has scoring and severity ratings, the short screen's primary use is as a binary screener (presence/absence of risk).
Adverse events | Days 1, 7, 14, 30, 90 post-block
  The occurrence of adverse events will be collected.
Sleep and Dream Log | Daily starting from 2 weeks before the block and ending at 2 weeks post-block
  A self-reported daily diary in which participants record details about their sleep patterns and dream experiences. Typical entries include bedtime, wake time, sleep latency, number and duration of awakenings, subjective sleep quality, and dream recall or content. The log provides qualitative and quantitative data on sleep behavior and dream activity over the monitoring period.
Daily Mood Questionnaire | Daily starting from 2 weeks before the block and ending at 2 weeks post-block
  A brief self-report instrument completed daily to assess fluctuations in mood states. Participants rate their current mood or specific affective dimensions (e.g., happiness, sadness, anxiety, irritability) using Likert-type scales. The questionnaire captures short-term mood variability and overall emotional well-being throughout the study period.
Home Sleep Monitoring | Daily starting from 2 weeks before the block and ending at 2 weeks post-block
  Objective sleep data collected at home using the Muse EEG headband, a wearable device that records brainwave activity to assess sleep architecture and quality. The device measures parameters such as sleep onset latency, total sleep time, sleep stages (e.g., REM, deep sleep), and awakenings. Data are analyzed to provide quantitative metrics of sleep patterns in a naturalistic environment.
Home-Based Polysomnography (PSG) | Three days before the block and 3 days post-block
  Participants will come to the lab in the evening, where study staff will attach a portable PSG device. Participants will then return home via taxi and sleep while wearing the device. The next morning, they will return to the lab via taxi, where the study staff will remove the PSG.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Liu Y, Li H, Hu Y, Yu S, Liu Q, Chen Y. Stellate Ganglion Block Improves Postoperative Cognitive Dysfunction in aged rats by SIRT1-mediated White Matter Lesion Repair. Neurochem Res. 2022 Dec;47(12):3838-3853. doi: 10.1007/s11064-022-03800-z. Epub 2022 Oct 31. PMID 36315371
- [Background] Yu K, Zhang XK, Xiong HC, Liang SS, Lu ZY, Wu YQ, Chen Y, Xiao SJ. Stellate ganglion block alleviates postoperative cognitive dysfunction via inhibiting TLR4/NF-kappaB signaling pathway. Neurosci Lett. 2023 Jun 11;807:137259. doi: 10.1016/j.neulet.2023.137259. Epub 2023 Apr 17. PMID 37075883